CLINICAL TRIAL: NCT03377413
Title: Novel Equation for Estimating Resting Energy(REE) Expenditure in Chronic Kidney Disease(CKD) 3-5 Stages Patients
Brief Title: Novel Equation for Estimating Resting Energy Expenditure
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong Jie, Clinical Professor in Renal Division, Department of Medicine, Peking University First Hospital
Other Study IDs: REE equation
Record Dates: First submitted 2017-12-14; First posted 2017-12-19 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Resting Energy Expenditure; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The energy and nutrition states are closely associated with CKD patients complications and outcomes.To reach the energy balance target, we need the accurate resting energy expenditure level of patients. Traditional equations are not applicable to CKD patients,so we aim to develop and validate a equation for estimating resting energy expenditure in CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* CKD 3-5 stages
* Age:18-80 years old

Exclusion Criteria:

* Dialysis and kidney transplantation;
* Acute complications to hospitalization
* 1 month prior to the study;
* Acute or chronic infections, cancer and other wasting diseases in the past year;
* Thyroid dysfunction;
* Acute onset of podagra; Musculoskeletal diseases;
* Respiratory diseases (asthma, pleural effusion, pneumothorax, COPD);
* History of hormonal drugs use;
* During pregnancy or lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic kidney disease 3-5 stages
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Novel equation development | September 1, 2017 to June 1, 2018
  Developed equation for estimating REE in CKD 3-5 stages patients
Novel equation validation | June 1, 2018 to March 1, 2019
  Validate the noval equation with REE obtained by indirect calorimetry (IC).

CONTACTS AND LOCATIONS:
Overall Officials: Jie Dong, Study Director — Renal Division and Institute of Nephrology, Peking University First Hospital
Locations (1):
- Renal Division and Institute of Nephrology, Peking University First Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Xu X, Yang Z, Ma T, Li Z, Chen Y, Zheng Y, Dong J. Novel equation for estimating resting energy expenditure in patients with chronic kidney disease. Am J Clin Nutr. 2021 Jun 1;113(6):1647-1656. doi: 10.1093/ajcn/nqaa431. PMID 33693520